CLINICAL TRIAL: NCT01472263
Title: Effectiveness of Pentoxifylline in Attenuating Neurological Disease Associated With HTLV-1 and Negative Modulator of Pathological Immune Response.
Brief Title: Use of Pentoxifylline in Human T-lymphotropic Virus Type-1 (HTLV-1) Diseases
Acronym: Pentox
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Universitário Professor Edgard Santos (Other)
Responsible Party: Principal Investigator, Davi Tanajura Costa, MD, Hospital Universitário Professor Edgard Santos
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INCT-DT
Record Dates: First submitted 2011-11-11; First posted 2011-11-16 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: HTLV-1; Tropical Spastic Paraparesis; Immune System Diseases; Physical Disability; Pentoxifylline
Keywords: HTLV-1; tropical spastic paraparesis; Immune System Diseases; Physical disability; pentoxifylline
MeSH Terms: conditions — Paraparesis, Tropical Spastic; Immune System Diseases | interventions — Pentoxifylline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pentoxifylline (Experimental)
  Interventions: Drug: Pentoxifylline
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pentoxifylline — Pentoxifylline 400mg 3 times a day on a total dose o 1200mg, oral capsules
  Other Names: Trental
  Arms: Pentoxifylline
Drug: Placebo — Placebo capsules 3 times a day. The capsules have the same shape, color and form as the treatment group, and are identified by envelope numbers.
  Arms: Placebo

SUMMARY:
In this study the investigators are going to evaluate the efficacy pentoxifyline in HTLV-1 patients with neurological diseases: HAM/TSP or neurogenic bladder. In some laboratory experiments the investigators observed that this drug had the capacity to reduce the immune response in HTLV-1 infected cells. Since the exacerbated immune response is know to cause neurological disease in patients with HTLV-1 the investigators hope that pentoxifyline can alleviate symptoms and delay the progress of HAM/TSP in patients.

DETAILED DESCRIPTION:
The human T-lymphotropic virus type 1 (HTLV-1) infects 20 million individuals worldwide and is the causative agent of HTLV associated myelopathy/ tropical spastic paraparesis (HAM/TSP). Although only 5% of HTLV-infected individuals will develop HAM/TSP, the investigatorts have observed that about 30% have neurological complaints and/or neurogenic bladder associated with HTLV-1. The immunopathogenesis of those diseases is related to the exaggerated immune response with high production of cytokines and induced neurological injury. So far there is not any effective drug against HTLV-1 and modulation of the immune response can help to alleviate the clinical manifestations of those patients and prevent the progression of symptoms. The preliminary data show that pentoxifylline has ability to decrease production of TNF-α and IFN-γ in patients with HTLV-1 infection and patients with HAM/TSP. The proposal entitled "Evaluation of the efficacy of pentoxifylline in attenuating the neurological disease associated with HTLV-1 and negatively modulate the immune pathological response" extends the previous studies in order to determine the ability of pentoxifylline in modulate the immune response and modify the course of the clinical manifestations in patients infected with HTLV-1. The influence on the immune response in the expression of disease will be determined in a therapeutic trial with two groups of patients: 1) patients with neurogenic bladder associated with HTLV-1, 2) patients with HAM/TSP. Primary end point is clinical and neurological exam and secondary end point are measure of proinflammatory cytokines (TNF-α, IFN-γ, IL-1 and IL-6) and chemokines that attract T cells to sites of inflammation (CXCL9 and CXCL10).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 80 years;
* Confirmed HTLV-1 infection with Western Blot analysis;
* HAM/TSP diagnosed patients according to the WHO
* Patients with HTLV-1 and neurogenic bladder diagnosed by clinical and urodynamic study
* Disease duration < 5 years

Exclusion Criteria:

* Neurological diseases with functional limitations.
* Co-infection with Hepatitis B or C, Syphilis, Chagas Disease or HIV
* Use of immunossupressive drugs
* Immune disease
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2009-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Functional neurological capacity | 60 days
  Measure of functional neurological capacity with the Expanded Disability Status Scale (EDSS), OSAME Motor Disability Score and Ambulatorial index

SECONDARY OUTCOMES:
Reduce in cytokines and chemokines | 60 days
  Measure of reduce in inflammatory cytokines (TNF alpha, IFN gamma, IL10 and IL5) and chemokines (CXCL9 and CXCL10)

CONTACTS AND LOCATIONS:
Overall Officials: Davi Costa, MD, Principal Investigator — Federal University of Bahia; André Muniz Santos, MD, PhD, Study Director — Federal University of Bahia; Edgar M Carvalho, MD, PhD, Study Chair — Federal University of Bahia
Locations (1):
- Hospital Universitário Professor Edgard Santos, Salvador, Estado de Bahia, Brazil